CLINICAL TRIAL: NCT06684704
Title: Comparison of Intraocular Pressure (Icare Non-contact Tonometry), Optic Nerve Sheath Diameter and Optic Perfusion Pressure of Minimal Low and High-Flow Anesthesia in Percutaneous Nephrolithotomy (Randomized, Prospective, Clinical Study)
Brief Title: Intraocular Pressure, Optic Nerve Sheath Diameter and Optic Perfusion Pressure of Minimal Low and High-Flow Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: FSCH-SB-2024/09-46
Record Dates: First submitted 2024-11-09; First posted 2024-11-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia; Intraocular Pressure; Nephrolithiasis
Keywords: Minimal Low-Flow Anesthesia; Percutaneous Nephrolithotomy; Optic Nerve Sheath Diameter; non-contact tonometry
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participants and investigators were blinded to the treatment assignments. The study utilized identical appearing interventions to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Low-Flo Anesthesia (Other): Group M minimal flow (n=30, fresh gas flow 0.5 L/min)
  Interventions: Other: minimal and high flow anesthesia
- High-Flow Anesthesia (Other): Group Y high flow (n=30, fresh gas flow 4 L/min).
  Interventions: Other: minimal and high flow anesthesia

INTERVENTIONS:
Other: minimal and high flow anesthesia — Low-flow anesthesia technique is a technique based on the re-breathing of at least half of the gas exhaled in semi-closed systems by returning at least half of the exhaled gas to the patient in the next inspiration.

SUMMARY:
The aim of this clinical trial is to determine the effect of minimal low-flow versus high-flow anesthesia on intraocular pressure (IOP) by non-contact tonometry, optic nerve sheath diameter (ONSD) by USG and optic perfusion pressure (OPP) in percutaneous nephrolithotomy operations. He will also learn about the effect on hemodynamic responses and arterial oxygenation. The main questions it aims to answer are:

What are the effects of low-flow anesthesia combined with prone position on intraocular pressure (IOP), optic nerve sheath diameter (ONSD) and optic perfusion pressure (OPP)? Which anesthesia flow type has optimal eye-protective results? The investigators will compare minimal low-flow and high-flow anesthesia.

Participants:

The study will include patients between the ages of 18-60 years with ASA (American Society of Anesthesiologists) risk classification I-II-III, who are scheduled for unilateral percutaneous nephrolithotomy (PCNL) operation in the Urology Clinic under elective conditions and who have given informed consent.

DETAILED DESCRIPTION:
Today, rapidly depleting resources and deteriorating ecosystems bring the concept of sustainability to the forefront in all areas. Anesthesia applications have also become an important evaluation subject in terms of sustainability. One of the important components of sustainable anesthesia is low-flow anesthesia. Low-flow anesthesia technique is a technique based on the re-breathing of at least half of the gas exhaled in semi-closed systems by returning at least half of the exhaled gas to the patient in the next inspiration (1). This reduces anesthetic gas consumption, reduces the carbon footprint and prevents environmental pollution. In addition, low-flow anesthesia protects mucociliary clearance mechanisms by preventing airway moisture loss and supports the physiological balance of the respiratory system (2). With the widespread use of low-flow anesthesia, research on the systemic effects of this method compared to high-flow anesthesia has also increased. Prone position may lead to undesirable effects such as increased intracranial pressure, increased intraocular pressure, increased cerebral blood flow and atelectasis. Although the effects of this position on intracranial and intraocular pressure are well known, studies on the effect of low-flow anesthesia on these parameters are limited. Therefore, how the use of low-flow anesthesia in combination with the prone position changes these effects should be evaluated in larger-scale studies (3).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60 years
* ASA (American Society of Anesthesiologists) risk classification I-II-III
* Unilateral percutaneous nephrolithotomy (PCNL) operation

Exclusion Criteria:

* Patients with drug and alcohol addiction,
* long-term smoking history (at least 1 pack/1 year),
* BMI>35,
* chronic lung disease,
* cerebrovascular disease,
* severe systemic diseases such as kidney, liver or advanced heart failure .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (ONSD) measurements | Measurements will be performed serially after induction of anesthesia (T0), 1 min after intubation (T1), 30 min after supine position (T2), supine from prone position (T3) and 5 min after extubation (T4).
  ONSD measurement bedside ultrasonography (POCUS) will be performed in accordance with the standardized ONSD POCUS Quality Criteria Checklist (ONSD POCUS QCC)

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | Measurements will be performed serially after induction of anesthesia (T0), 1 min after intubation (T1), 30 min after supine position (T2), supine from prone position (T3) and 5 min after extubation (T4).
  Intraocular pressure (IOP) is calculated by spraying air into the center of the cornea with a noncontact tonometer and measuring the reflected air again by slightly flattening the cornea.

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Seçiniz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jang YE, Nam S, Ji SH, Kim EH, Lee JH, Jung JH, Kim HS, Kim JT. Effect of end-tidal carbon dioxide level on the optic nerve sheath diameter measured by transorbital ultrasonography in anesthetized pediatric patients: A randomized trial. Paediatr Anaesth. 2022 Jun;32(6):754-763. doi: 10.1111/pan.14437. Epub 2022 Mar 20. PMID 35279906
- [Background] Mermer A, Kozanhan B. Comparison of the effects of low-flow and normal-flow anesthesia on intracranial pressure, cerebral oxygenation and bispectral index in laparoscopic cholecystectomy operation. Eur Rev Med Pharmacol Sci. 2023 Sep;27(18):8514-8522. doi: 10.26355/eurrev_202309_33776. PMID 37782167